CLINICAL TRIAL: NCT04393350
Title: WINSHIP4955-20: Perioperative Lenvatinib With Pembrolizumab in Patients With Locally Advanced Nonmetastatic Clear Cell Renal Cell Carcinoma
Brief Title: Perioperative Lenvatinib With Pembrolizumab in Patients With Locally Advanced Nonmetastatic Clear Cell Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mehmet Bilen, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000009; NCI-2020-01064 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4955-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Kidney Cancer; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (lenvatinib, pembrolizumab) (Experimental): Patients receive lenvatinib PO QD on days 1-21 and pembrolizumab IV over 30 minutes on day 1. Treatments repeat every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenvatinib; Drug: Lenvatinib Mesylate; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Lenvatinib — Given PO
  Other Names: E7080; ER-203492-00; Multi-Kinase Inhibitor E7080
Drug: Lenvatinib Mesylate — Given PO
  Other Names: 4-[3-Chloro-4-(N''-cyclopropylureido)phenoxy]7-methoxyquinoline-6-carboxamide Mesylate; E7080; Lenvima; Multi-Kinase Inhibitor E7080
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well lenvatinib and pembrolizumab before surgery work in treating patients with kidney cancer that has spread from its original site of growth to nearby tissues or lymph nodes but has not spread to other places in the body (non-metastatic). Lenvatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving lenvatinib and pembrolizumab before surgery may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the objective response rate (complete and partial responses), following the administration of lenvatinib and pembrolizumab for a total of 4 cycles (12 weeks) in patients with locally-advanced, biopsy-proven non-metastatic clear cell renal cell carcinoma (ccRCC) prior to undergoing nephrectomy (partial or radical).

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of neoadjuvant lenvatinib plus pembrolizumab in a presurgical population as well as the safety of adjuvant pembrolizumab post-surgery.

II. To determine the clinical outcomes including disease-free survival (DFS) and overall survival (OS) of patients with non-metastatic ccRCC treated with neoadjuvant lenvatinib and pembrolizumab and adjuvant pembrolizumab.

III. To evaluate surgery-related complications and outcomes as per the Clavien-Dindo classification system.

EXPLORATORY OBJECTIVES:

I. To evaluate changes in biomarkers of immune activation and gene expression before, during and after treatment.

II. To assess the quality of life, frailty and sarcopenia of patients before and after treatment.

OUTLINE:

Patients receive lenvatinib orally (PO) once daily (QD) on days 1-21 and pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatments repeat every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 14 days, then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a renal mass consistent with a clinical stage >= T3Nx or TanyN+ or deemed unresectable by surgeon
* Renal cell carcinoma with clear cell component on pre-treatment biopsy of the primary tumor
* The participant (or legally acceptable representative if applicable) provides written informed consent and the willingness and ability to comply with all aspects of the protocol
* Have an Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Absolute neutrophil count (ANC) >= 1500/uL (specimens must be collected within 72 hours prior to the start of study treatment)
* Platelets >= 100 000/uL (specimens must be collected within 72 hours prior to the start of study treatment)
* Hemoglobin >= 9.0 g/dL (specimens must be collected within 72 hours prior to the start of study treatment) or ≥5.6 mmol/La

Renal:

Creatinine =≤1.5 × ULN OR Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl)=≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN.

Hepatic:

Total bilirubin=≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN AST (SGOT) and ALT (SGPT)=≤2.5 × ULN (≤5 × ULN for participants with liver metastases)

Coagulation:

International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT)=≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.

ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

* Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
* Creatinine clearance (CrCl) should be calculated per institutional standard.

  * International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x upper limit of normal (ULN) unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants (specimens must be collected within 72 hours prior to the start of study treatment)
  * Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (specimens must be collected within 72 hours prior to the start of study treatment)
  * Serum creatinine =< 1.5 x ULN OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 40 mL/min (>= 0.67 mL/sec) for participant with creatinine levels > 1.5 x institutional ULN (specimens must be collected within 72 hours prior to the start of study treatment)
* Creatinine clearance (CrCl) calculated per the Cockcroft and Gault formula

  * Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (specimens must be collected within 72 hours prior to the start of study treatment)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN (=< 5 x ULN for participants with liver metastases) (specimens must be collected within 72 hours prior to the start of study treatment)
  * All females must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of beta-human chorionic gonadotropin [beta-hCG]) at the screening visit and the baseline visit. A pregnancy test needs to be performed within 72 hours of the first dose of study drug. Women of childbearing potential (WOCBP) must agree to use a highly effective method of contraception for the entire study period and for 120 days after study discontinuation
  * Male subjects who are partners of women of childbearing potential must use a condom and their female partners of childbearing potential must use a highly effective method of contraception beginning at least 1 menstrual cycle prior to starting study drugs, throughout the entire study period, and for 120 days after the last dose of study drug, unless the male subjects are totally sexually abstinent or have undergone a successful vasectomy with confirmed azoospermia or unless the female partners have been sterilized surgically or are otherwise proven sterile

Exclusion Criteria:

* Evidence of metastatic disease on pre-treatment imaging
* The subject has received of any type of cytotoxic, biologic or other systemic anticancer therapy for kidney cancer
* The subject has received any other type of investigational agent within 28 days before the first dose of study treatment
* Excluding the primary tumor leading to enrollment in this study, any other active malignancy (except for localized prostate cancer, definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the bladder or cervix) within the past 24 months
* Prior treatment with lenvatinib or any agent directed against PD-1, PD-L1 or PD-L2, or another stimulatory or co inhibitory T-cell receptor (e.g. CTLA-4, OX 40, CD137)
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment
* Subjects having > 1+ proteinuria on urinalysis will undergo 24-hour urine collection for quantitative assessment of proteinuria. Subjects with urine protein >= 1 g/24-hour will be ineligible
* Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * New York Heart Association congestive heart failure of grade II or above, unstable angina, myocardial infarction within the past 6 months, or serious cardiac arrhythmia associated with significant cardiovascular impairment within the past 6 months
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment
    * Prolongation of corrected QT (QTc) interval to > 480 msec per electrocardiogram (ECG) within 28 days before first dose of study treatment
  * Clinically significant hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g. pulmonary hemorrhage) within 3 weeks prior to the first dose of study drug
  * Serious non-healing wound/ulcer/bone fracture
  * History of organ allograft (subject has had an allogenic tissue/solid organ transplant)
* Biologic response modifiers (e.g. granulocyte colony-stimulating factor) within 4 weeks before study entry. Chronic erythropoietin therapy is permitted provided that no dose adjustments were made within 2 months before first dose of study treatment
* Subjects must have recovered adequately from any toxicity and/or complications from major surgery prior to starting therapy
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist are live attenuated vaccines and are not allowed
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of active Hepatitis B (e.g., hepatitis B surface antigen [HBsAg]) or hepatitis C (e.g., HCV RNA qualitative is detected)
* Has uncontrolled HIV defined by a CD4+ count < 350 cells/uL, an AIDS-defining opportunistic infection within the last 12 months prior to study enrollment or documented multidrug resistance that prevents effective HIV therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (complete and partial responses) | Baseline until end of Cycle 1 (4 Cycles (12 weeks)
  Will assess the proportion of patients with a reduction in overall tumor burden from baseline after 12 weeks of treatment with neoadjuvant lenvatinib and pembrolizumab.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | From treatment phase up to 14 day post treatment
  Adverse events will be assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The safety profile of the treatment will be documented and summarized by summary statistics as frequency and percentage for each AE.
Overall survival (OS) | Up to 4 years after study start
  OS will be estimated with the Kaplan-Meier method. The OS of each patient group at specific time points such as 6 months, 1 year, 3 years, etc. and will be also estimated alone with 95% confidence interval (CI).
Disease free survival (DFS) | From time of surgery to the first tumor recurrence, or death, assessed up to 4 years
  DFS will be estimated with the Kaplan-Meier method. The DFS of each patient group at specific time points such as 6 months, 1 year, 3 years, etc. and will be also estimated alone with 95% CI.

OTHER OUTCOMES:
Biomarker analysis | Up to 4 years after study start
  Paired t-test or Wilcoxon singed-rank test will be used to compare the biomarkers change before, during, and after treatment.
Quality of life: Functional Assessment of Cancer Therapy-Kidney Specific Index-19 questionnaire | Up to 4 years after study start
  QOL will be assessed using the Functional Assessment of Cancer Therapy-Kidney Specific Index-19 (FKSI-19) questionnaire. Summary statistics will be applied to all items in the measurements for quality of life. The KSI-19 is an experimental end point. The minimum and maximum values and whether higher scores mean a better or worse outcome will be determined once data is collected.
Fried Frailty Score | Up to 4 years after study start
  Will be assessed using the using the Fried Frailty score. Summary statistics will be applied to all items in the measurements for frailty. The Fried Frailty Score is an experimental end point. The minimum and maximum values and whether higher scores mean a better or worse outcome will be determined once data is collected.
Degree of sarcopenia | Up to 4 years after study start
  Will assess pre-and post-treatment imaging via SliceOmatic version (V) 5.0 by TomoVision program. Summary statistics will be applied to all items in the measurements for degree of sarcopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet A Bilen, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Results of the trial and not individual patient data will be shared. The study protocol, consent, and investigator's brochure will be available. The statistical plan is incorporated into the protocol, along with inclusion and exclusion criteria.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT04393350/Prot_SAP_000.pdf